CLINICAL TRIAL: NCT07059325
Title: Accelerated, Left Prefrontal Transcranial Magnetic Stimulation for Functional Seizures; An Open-Label Exploration of Feasibility, Tolerability, and Preliminary Efficacy
Brief Title: Accelerated TMS for Seizure-Type Functional Neurologic Disorders
Acronym: FND-seiz
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Joseph Chasen, Principle Investigator, Resident Physician, MUSC Departments of Psychiatry and Neurology, Medical University of South Carolina
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00144502
Record Dates: First submitted 2025-06-16; First posted 2025-07-10 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Functional Neurological Symptom Disorder; Functional Seizures
Keywords: Mental Health; Psychiatry; Functional Seizures; Transcranial Magnetic Stimulation
MeSH Terms: conditions — Conversion Disorder; Psychogenic Nonepileptic Seizures; Psychological Well-Being | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: This is a single-arm open label investigation of the safety, feasibility, and tolerability of an accelerated TMS protocol in patients with Functional Seizures, also known as Psychogenic Non-Epileptic Seizures, with a secondary aim of examining preliminary efficacy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Interventional Arm (Experimental)
  Interventions: Device: Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation — Participants will receive 6 to 10 sessions per day (i.e., theta burst; 600 pulses per session; 6000 pulses per day) over 3 to 5 treatment days using a MagVenture MagPro TMS System. Treatment will consist of a total of 30 sessions (18,000 total pulses). A single session is defined as 600 pulses at 50 Hz for 2s (i.e., 5 Hz triplets) and repeated every 10s for a total of 190s per session to l-dlPFC at 120% rMT with 15-minute intersession intervals. TMS will be targeted to Beam F3 for comparison to the bulk of the literature and to most mimic replicable clinical use.
  Other Names: Accelerated TMS; Theta-burst TMS

SUMMARY:
The purpose of this project is to assess the feasibility, tolerability, and preliminary efficacy of using an accelerated, intermittent theta burst stimulation (a-iTBS-rTMS) protocol targeting the left dorsolateral prefrontal cortex (l-dlPFC) for Psychogenic Non-Epileptic Seizures (PNES) or Seizure-Type Functional Neurologic Disorder (FND-seiz) in an open-label fashion. Following screening, consent, and enrollment, participants will receive 6-to-10 iTBS-rTMS sessions per day (i.e., theta burst; 600 pulses per session; 6000 pulses per day) over a 3-to-5 treatment days with a target of 30 total sessions (18,000 total pulses). TMS will be targeted to Beam F3 for comparison to the bulk of the literature and to most mimic replicable and clinical use. This proposed iTBS-rTMS protocol was chosen given its previously shown safety, tolerability, and effectiveness in other conditions, but also as it has the potential to shorten treatment to only 3 days, which investigators theorize will be more feasible for patients with FND-seiz.

Feasibility will be measured as the percentage of participants who receive at least 20 treatment sessions within the 3-to-5-day window. Other than self-assessments used in the safety screening process or to monitor TMS benefits and risks, secondary subjective measures will assess previously investigated FND-seiz-specific outcomes, which will be obtained prior to intervention and 4-weeks post-intervention. In addition to monthly seizure frequency, this will include validated measures regarding stigma, health-related QOL, depression, PTSD, somatic symptoms, psychosocial functioning, psychological distress, and clinical and participant impression of improvement and satisfaction. Sub-analysis will further divide participants with mild to no depression and/or PTSD versus moderate to severe depression and/or PTSD to further assess how the TMS effects known to effect other highly comorbid disorders with FND-seiz, may indirectly affect FND-seiz outcomes.

DETAILED DESCRIPTION:
Seizure-Type Functional Neurologic Disorders (FND-seiz) are strikingly prevalent-accounting for 5-15% of epilepsy center referrals and up to 40% of epilepsy monitoring unit admissions-when considering the associated barriers to treatment and dismal outcomes. Due to resource-intensive requirements, diagnosis is often delayed by years. In the interim, patients frequently receive inappropriate antiseizure medications and have high utilization of emergency services. Years after diagnosis, many FND-seiz patients continue to experience non-epileptic seizures (NS) and have high rates of disability. Due to stigma and psychosocial barriers, engagement and responses to the standard of care, Cognitive Behavioral Therapy (CBT), are inconsistent. As many patients are told they may have epilepsy prior to receiving an accurate diagnosis, there is an obvious disconnect between the recommended psychological treatment and the physical nature of their symptoms, which can limit acceptance of the diagnosis and subsequently CBT engagement. Furthermore, the only powered RCT (the CODES trial) examining CBT in FND-seiz failed to show a significant seizure reduction at 12 months follow up and the overall effect size was lower than previously thought highlighting the limitations of a "one-size-fits-all" model for a highly comorbid disorder. Ultimately, patients with FND-seiz have been found to have a poorer overall quality of life compared to epilepsy and a standardized mortality rate 2.5 times greater the general population and comparable to that of drug-resistant epilepsy

Together these factors underscore the need for alternate treatments capable of addressing psychosocial challenges unique to FND-seiz or further investigating the underlying neurobiology. Investigators theorize that offering a brain-network based approach may reduce stigma associated with confusion over the "psychological" rather than "neurological" etiologic conception of FND-seiz, which if effective, may be a more feasible for some patients. Brain-imaging research and prior reports of benefit with neurostimulation suggests TMS to the left dorsolateral prefrontal cortex (l-dlPFC) has the potential to improve cortico-limbic or cortico-sensorimotor governance, which Investigators theorize in FND-seiz may decrease NS frequency or improve quality of life. Thus, Investigators aim to investigate the feasibility and tolerability of an accelerated, intermittent theta-burst TMS protocol in FND-seiz to best mimic current clinical trends and optimize TMS feasibility, which may have several applications for the FND-seiz population.

In clinical practice, the known, but rare risk of inducing an epileptic seizure with TMS and the difficulty differentiating epileptic from non-epileptic seizures, may decrease the comfort of TMS providers to use TMS in FND-seiz patients when indicated for other disabling disorders. In tandem with exploring the feasibility and tolerability of this intervention, Investigators hope to employ and investigate an informed safety protocol, with input from experts in the fields of epilepsy and brain stimulation. Helping providers safely screen patients, more decisively exclude patients with an inaccurate diagnosis or concomitant epilepsy and having a protocol to follow when treating FND-seiz patients who experience a NS during TMS stimulation may increase TMS access for FND-seiz patients with other TMS indications. Finally, as preliminary evidence here at MUSC also suggests combining TMS with CBT for other indications may have a synergistic effect and improve attrition with CBT, if TMS is preliminarily efficacious alone in FND-seiz specific outcomes in a small, open-label sample, this investigation may also help optimize future methodologies examining the use of TMS in FND-seiz.

ELIGIBILITY:
Inclusion Criteria:

1. >18 years old and <65 years old
2. English Speaking, can read and write, and able to provide informed consent
3. Diagnosis of "documented" Functional Seizures as made by an MUSC epileptologist or neurologist using the ILAE recommendations: "by clinician experienced in diagnosis of seizure disorders (on video or in person), showing semiology of typical of FND-seiz, while on EEG plus no epileptiform activity on routine or ambulatory ictal EEG during a typical ictus/event in which the semiology would make ictal epileptiform EEG activity expected during equivalent epileptic seizures"2
4. In addition to meeting ILAE minimum requirements for FND-seiz diagnosis, must have previously undergone and documented in the electronic medical record a minimum of 24-hours of otherwise normal video EEG without interictal epileptiform findings
5. Duration of symptoms >3 months and continuing to experience NES at least monthly
6. Not currently undergoing any psychotherapeutic intervention, agree to forgo any psychotherapeutic intervention during the study, and if previously completed any psychotherapeutic intervention continue to experience monthly non-epileptic seizures
7. If on psychotropic medications may choose to continue during the duration of the study at current doses, but consent to not modifying medication doses or switching to alternative psychotropic regimens during the trial
8. In good general health, as ascertained by medical history
9. Females of reproductive age (ages 18 to 50) must have a negative urine pregnancy test, performed onsite, and documented in the study record within 72 hours prior to the first TMS session

Exclusion Criteria:

1. History of clinical concern for concomitant epileptic seizures or epilepsy
2. History of ongoing psychosis, mania, active alcohol or substance use disorder as screened by the PSQ, YMRS, AUDIT, and DAST-10
3. History of positive screening urine test for drugs of abuse within the last year: cocaine, amphetamines, barbiturates, opiates
4. Active suicidal intent or a score >2 on question 3 of the HAM-D
5. Use of medications known to lower the seizure threshold at doses that may increase this risk in the setting of rTMS-iTBS (i.e. buproprion at >300 mg, combinations of tricyclic antidepressants, antipsychotics… as determined by investigators)
6. History of central nervous system surgeries or clinically relevant structural brain lesions
7. Significant or unstable cardiac, metabolic, oncologic, psychiatric, developmental, or neurologic condition(s) or treatments that may impact safe participation in the study as determined by the study investigators (e.g. poorly-controlled heart failure, current or past cardiac arrhythmia, sustained systolic blood pressure >180, labile diabetes, significant electrolyte abnormality, brain cancer, cognitive impairment, neurodevelopmental disorders, autism spectrum disorder, mania, schizophrenia spectrum or other psychotic disorder, movement disorders, multiple sclerosis, moderate to severe brain injury)
8. Participation in any clinical trial with an investigational drug or device within the past month or concurrent to study participation
9. History of TMS exposure
10. TMS contraindications (e.g., ferromagnetic implants, cochlear implants, conditions or treat-ments that lower seizure threshold - as determined by study investigators).
11. Current pregnancy or desire to become pregnant during study duration without contraceptive plan
12. Are a prisoner or in police custody at the time of eligibility screening

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-09-02 (Actual); Primary Completion 2026-09-02 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Completing TMS Sessions | Assessed daily from Day 1 to Day 5 of the TMS treatment period and summarized at the 4-week follow-up visit.
  Description: Feasibility will be measured as the percentage of participants who complete at least 20 rTMS-iTBS treatment sessions within the 3-to-5-day treatment period.
  Unit of Measure: Percentage (%) Time Frame: Assessed daily from Day 1 to Day 5 of the TMS treatment period and summarized at the 4-week follow-up visit.
  Rationale: This measure focuses on the proportion of participants able to adhere to the intensive TMS protocol, a key indicator of feasibility. The time frame is now specific, covering the treatment days (Day 1 to Day 5) and the 4-week follow-up for final reporting.
Session Delivery Patterns | Recorded daily from Day 1 to Day 5 of the TMS treatment period and summarized at the 4-week follow-up visit.
  Description: The number of total rTMS-iTBS sessions delivered will be recorded and analyzed to characterize protocol adherence and delivery patterns. rTMS-iTBS sessions within the protocol are aimed to be delivered over the 3-5 treatment days, during which participants may choose between 6-10 day treatment sessions per day if tolerable and feasible (total of 30 sessions to complete the rTMS-iTBS protocol) Unit of Measure: The number of sessions delivered, represented as a continuous, numerical value.
  Rationale: This measure provides additional detail on how the protocol is implemented, addressing potential variability in session delivery to assess overall tolerability, feasibility, and analyze any potential adverse events. It further helps inform measures of efficacy if participants do not complete the total session target or complete the course of different time periods (ie, over 4-5 days or over 3 days).
Adverse Event Rate | Assessed daily from Day 1 to Day 5 of the TMS treatment period, at the initial screening visit (baseline), and at the 4-week follow-up visit.
  Description: Tolerability will be assessed by calculating the percentage of participants experiencing at least one adverse event (AE) related to the rTMS-iTBS protocol, such as headache, scalp discomfort, or dizziness. Adverse events will be recorded and classified using a standardized checklist based on common TMS-related side effects.
  Unit of Measure: Percentage (%) of participants with at least one AE. Rationale: This measure quantifies the proportion of participants experiencing AEs, providing a clear indicator of the protocol's tolerability. Daily assessments during treatment capture immediate side effects, while the 4-week follow-up evaluates any delayed or persistent effects.
Serious Adverse Event Rate | Assessed daily from Day 1 to Day 5 of the TMS treatment period, at the initial screening visit (baseline), and at the 4-week follow-up visit.
  Description: Serious adverse events (SAEs), defined as any event resulting in hospitalization, life-threatening conditions, or significant disability (e.g., seizure), will be tracked and reported as the percentage of participants experiencing at least one SAE related to the rTMS-iTBS protocol.
  Unit of Measure: Percentage (%) of participants with at least one SAE. Rationale: This measure ensures monitoring of severe outcomes, which is critical for assessing the safety of the TMS protocol. The specific time points align with the study's schedule, ensuring comprehensive tracking of rare but serious events.
Pulses per Session Delivery Patterns | Recorded daily from Day 1 to Day 5 of the TMS treatment period and summarized at the 4-week follow-up visit.
  Description: The number and frequency of rTMS-iTBS pulses delivered over the 3-5 treatment days during which participants may choose between 6-10 day treatment sessions per day. This will be recorded and analyzed to characterize protocol adherence and delivery patterns. A pulse is defined as a burst of three magnetic pulses delivered in quick succession. One treatment session entails 190s encompassing 600 pulses per session. An intermittent theta-burst pulse is defined as a burst of three magnetic pulses delivered in quick succession. The end point of 30 treatment sessions is 18,000 total pulses delivered, which over the 3 to 5 day window can be achieved with 3,600 daily pulses for 5 days or up to 6,000 daily pulses over 3 days.
  Unit of Measure: The number of sessions delivered, represented as a continuous, numerical value.
  Rationale: This measure provides additional detail on how the protocol is implemented, addressing potential variability in session delivery to assess overall tole

SECONDARY OUTCOMES:
Non-epileptic Seizure Frequency (NES) | Assessed prior to intervention at visit 1, 2-4 weeks prior to starting the 3-5 day TMS treatment protocol, and at the final follow up visit 4 weeks after completing the TMS treatment protocol.
  Participants will receive in-person and written documentation on how to document NES frequency (the number NES events over a 4 week period) following events ideally in tandem with a family or support persons who may live with them. The subject and their support person will be asked to document NES semiology, duration, and symptom severity to ensure the events in question are consistent with their known events that have been previously confirmed to represent NES with video EEG. Final analysis will represent a continuous variable comparing the numerical value (number of NES events over a 4 week period).
Chronic Illness Anticipated Stigma Scale (CIASS) | Assessed at initial visit (time point 0 at visit 1, 2-4 weeks pre-TMS) and at post-intervention follow-up (4 weeks post-TMS).
  Purpose: Measures anticipated stigma related to chronic illness in participants with functional seizures.
  Unit of Measure: Total score on a scale. Score Range: 12-60 (12 items, each scored 1-5). Type of Variable: Continuous (sum of item scores). Interpretation: Higher scores indicate greater anticipated stigma (worse outcome).
Montgomery-Asberg Depression Rating Scale (MADRS) | Assessed at initial visit (2-4 weeks pre-TMS) and follow-up (4 weeks post-TMS).
  Purpose: Assesses depression severity in participants with functional seizures. Unit of Measure: Total score on a scale. Score Range: 0-60 (10 items, each scored 0-6). Type of Variable: Continuous (sum of item scores). Interpretation: Higher scores indicate greater depression severity (worse outcome).
  Sub-analysis: Participants divided into mild/no depression (MADRS ≤ 20) vs. moderate/severe depression (MADRS > 20) to compare with FND-seizure-specific outcomes (e.g., NHS3, NES remission).
Post-Traumatic Stress Disorder Checklist for DSM-5 (PCL-5) | Assessed at initial visit (2-4 weeks pre-TMS) and follow-up (4 weeks post-TMS).
  Purpose: Evaluates PTSD symptom severity in participants with functional seizures.
  Unit of Measure: Total score on a scale. Score Range: 0-80 (20 items, each scored 0-4). Type of Variable: Continuous (sum of item scores). Interpretation: Higher scores indicate greater PTSD symptom severity (worse outcome).
  Sub-analysis: Participants divided into mild/no depression (MADRS ≤ 20) vs. moderate/severe depression (MADRS > 20) and absent/mild PTSD (PCL-5 < 33) vs. moderate/extreme PTSD (PCL-5 ≥ 33) to compare with FND-seizure-specific outcomes.
PROMIS®-29+2 Profile v2.1 (PROPr) | Assessed at initial visit (2-4 weeks pre-TMS) and follow-up (4 weeks post-TMS).
  Purpose: Measures health-related quality of life across multiple domains (physical function, anxiety, depression, fatigue, sleep disturbance, social function, pain intensity, pain interference).
  Unit of Measure: T-scores for each domain. Score Range: T-scores (mean = 50, SD = 10) for each domain; typically ranges from 20-80 depending on the domain.
  Type of Variable: Continuous (T-scores per domain).
  Interpretation:
  Physical function and social function: Higher scores indicate better outcomes. Anxiety, depression, fatigue, sleep disturbance, pain intensity, pain interference: Higher scores indicate worse outcomes.
Patient Health Questionnaire-15 (PHQ-15) | Assessed at initial visit (2-4 weeks pre-TMS) and follow-up (4 weeks post-TMS).
  Purpose: Assesses somatic symptom severity in participants with functional seizures.
  Unit of Measure: Total score on a scale. Score Range: 0-30 (15 items, each scored 0-2). Type of Variable: Continuous (sum of item scores). Interpretation: Higher scores indicate greater somatic symptom severity (worse outcome).
Clinical Outcomes in Routine Evaluation (CORE-10) | Assessed at initial visit (2-4 weeks pre-TMS) and follow-up (4 weeks post-TMS).
  Purpose: Measures general psychological distress in participants with functional seizures.
  Unit of Measure: Total score on a scale. Score Range: 0-40 (10 items, each scored 0-4). Type of Variable: Continuous (sum of item scores). Interpretation: Higher scores indicate greater psychological distress (worse outcome).
Clinical Global Impression-Improvement and Severity (CGI-I and CGI-S) | Time Frame: CGI-S assessed at initial visit (2-4 weeks pre-TMS) and follow-up (4 weeks post-TMS); CGI-I assessed only at follow-up (4 weeks post-TMS).
  Purpose: Assesses clinical severity (CGI-S) and improvement (CGI-I) in participants' functional seizure condition.
  Unit of Measure: Rating on a scale.
  Score Range:
  CGI-S: 1-7 (1 = normal, not at all ill; 7 = extremely ill). CGI-I: 1-7 (1 = very much improved; 7 = very much worse). Type of Variable: Ordinal (discrete ratings).
  Interpretation:
  CGI-S: Higher scores indicate greater illness severity (worse outcome). CGI-I: Higher scores indicate less improvement or worsening (worse outcome).
The National Hospital Seizure Severity Scale (NHS3) | Assessed at initial visit (2-4 weeks pre-TMS) and follow-up (4 weeks post-TMS).
  Purpose: Measures seizure severity in participants with functional seizures. Unit of Measure: Total score on a scale. Score Range: 0-27 (based on seizure characteristics, e.g., frequency, duration, injury).
  Type of Variable: Continuous (sum of weighted items). Interpretation: Higher scores indicate greater seizure severity (worse outcome).
Participants with Complete NES Remission | Assessed at follow-up (4 weeks post-TMS).
  Purpose: Determines the proportion of participants achieving complete remission of non-epileptic seizures (NES).
  Unit of Measure: Percentage of participants with no NES events. Score Range: Binary (0% or 100% remission per participant). Type of Variable: Binary (remission achieved or not). Interpretation: Achieving remission (100%) is a better outcome.
Participants with >50% Reduction in NES Frequency | Assessed at follow-up (4 weeks post-TMS).
  Purpose: Measures the proportion of participants with a significant reduction (>50%) in non-epileptic seizure frequency.
  Unit of Measure: Percentage of participants achieving >50% reduction in NES frequency.
  Score Range: Binary (≥50% reduction or <50% reduction per participant). Type of Variable: Binary (reduction achieved or not). Interpretation: Achieving >50% reduction is a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Chasen, DO, Principal Investigator — Medical University of South Carolina
Locations (1):
- Institute of Psychiatry, Brain Stimulation Department, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No
Other than demographics and rates of psychiatric comorbidity seen across participants that may effect results, as this is a psychiatrically vulnerable population, no IPD is planned to be shared.

REFERENCES:
- [Background] Kan RLD, Padberg F, Giron CG, Lin TTZ, Zhang BBB, Brunoni AR, Kranz GS. Effects of repetitive transcranial magnetic stimulation of the left dorsolateral prefrontal cortex on symptom domains in neuropsychiatric disorders: a systematic review and cross-diagnostic meta-analysis. Lancet Psychiatry. 2023 Apr;10(4):252-259. doi: 10.1016/S2215-0366(23)00026-3. Epub 2023 Mar 7. PMID 36898403
- [Background] Wang Y, Gao H, Qi M. Left dorsolateral prefrontal cortex activation can accelerate stress recovery: A repetitive transcranial stimulation study. Psychophysiology. 2023 Oct;60(10):e14352. doi: 10.1111/psyp.14352. Epub 2023 May 23. PMID 37221649
- [Background] Philip NS, Barredo J, van 't Wout-Frank M, Tyrka AR, Price LH, Carpenter LL. Network Mechanisms of Clinical Response to Transcranial Magnetic Stimulation in Posttraumatic Stress Disorder and Major Depressive Disorder. Biol Psychiatry. 2018 Feb 1;83(3):263-272. doi: 10.1016/j.biopsych.2017.07.021. Epub 2017 Aug 8. PMID 28886760
- [Background] Hassa T, Sebastian A, Liepert J, Weiller C, Schmidt R, Tuscher O. Symptom-specific amygdala hyperactivity modulates motor control network in conversion disorder. Neuroimage Clin. 2017 Apr 27;15:143-150. doi: 10.1016/j.nicl.2017.04.004. eCollection 2017. PMID 28529870
- [Background] Maurer CW, LaFaver K, Ameli R, Epstein SA, Hallett M, Horovitz SG. Impaired self-agency in functional movement disorders: A resting-state fMRI study. Neurology. 2016 Aug 9;87(6):564-70. doi: 10.1212/WNL.0000000000002940. Epub 2016 Jul 6. PMID 27385746
- [Background] Mcsweeney M, Reuber M, Levita L. Neuroimaging studies in patients with psychogenic non-epileptic seizures: A systematic meta-review. Neuroimage Clin. 2017 Jul 27;16:210-221. doi: 10.1016/j.nicl.2017.07.025. eCollection 2017. PMID 28808618
- [Background] Perez DL, Dworetzky BA, Dickerson BC, Leung L, Cohn R, Baslet G, Silbersweig DA. An integrative neurocircuit perspective on psychogenic nonepileptic seizures and functional movement disorders: neural functional unawareness. Clin EEG Neurosci. 2015 Jan;46(1):4-15. doi: 10.1177/1550059414555905. Epub 2014 Nov 27. PMID 25432161
- [Background] Perez DL, Nicholson TR, Asadi-Pooya AA, Begue I, Butler M, Carson AJ, David AS, Deeley Q, Diez I, Edwards MJ, Espay AJ, Gelauff JM, Hallett M, Horovitz SG, Jungilligens J, Kanaan RAA, Tijssen MAJ, Kozlowska K, LaFaver K, LaFrance WC Jr, Lidstone SC, Marapin RS, Maurer CW, Modirrousta M, Reinders AATS, Sojka P, Staab JP, Stone J, Szaflarski JP, Aybek S. Neuroimaging in Functional Neurological Disorder: State of the Field and Research Agenda. Neuroimage Clin. 2021;30:102623. doi: 10.1016/j.nicl.2021.102623. Epub 2021 Mar 11. PMID 34215138
- [Background] Nightscales R, McCartney L, Auvrez C, Tao G, Barnard S, Malpas CB, Perucca P, McIntosh A, Chen Z, Sivathamboo S, Ignatiadis S, Jones S, Adams S, Cook MJ, Kwan P, Velakoulis D, D'Souza W, Berkovic SF, O'Brien TJ. Mortality in patients with psychogenic nonepileptic seizures. Neurology. 2020 Aug 11;95(6):e643-e652. doi: 10.1212/WNL.0000000000009855. Epub 2020 Jul 20. PMID 32690794
- [Background] McLoughlin C, McWhirter L, Pisegna K, Tijssen MAJ, Tak LM, Carson A, Stone J. Stigma in functional neurological disorder (FND) - A systematic review. Clin Psychol Rev. 2024 Aug;112:102460. doi: 10.1016/j.cpr.2024.102460. Epub 2024 Jun 13. PMID 38905960
- [Background] Robson C, Myers L, Pretorius C, Lian OS, Reuber M. Health related quality of life of people with non-epileptic seizures: The role of socio-demographic characteristics and stigma. Seizure. 2018 Feb;55:93-99. doi: 10.1016/j.seizure.2018.01.001. Epub 2018 Jan 12. PMID 29414141
- [Background] Samuels T, Pretorius C. Healthcare providers' perspectives on stigma when working with people with functional seizures. Seizure. 2023 Nov;112:121-127. doi: 10.1016/j.seizure.2023.10.002. Epub 2023 Oct 1. PMID 37820427
- [Background] Karterud HN, Otto Nakken K, Lossius MI, Tschamper M, Ingebrigtesen T, Henning O. Young people diagnosed with psychogenic nonepileptic seizures (PNES) years ago - How are they now? Epilepsy Behav. 2024 Aug;157:109874. doi: 10.1016/j.yebeh.2024.109874. Epub 2024 Jun 7. PMID 38851124
- [Background] Abi-Nahed R, Li J, Carlier J, Birca V, Berube AA, Nguyen DK. Outcome of psychogenic non-epileptic seizures following diagnosis in the epilepsy monitoring unit. Front Neurol. 2024 Feb 14;15:1363459. doi: 10.3389/fneur.2024.1363459. eCollection 2024. PMID 38419704
- [Background] Fettig M, El-Hage W, Klemina I, Biberon J, de Toffol B, Thiriaux A, Visseaux JF, Lemesle Martin M, Schwan R, Bechiri F, Cohn A, Meyer M, Maillard L, Hingray C. Adherence to mental health care and caregiver-patient relationship after diagnosis of psychogenic non-epileptic seizures: Longitudinal follow-up study. Seizure. 2020 Aug;80:227-233. doi: 10.1016/j.seizure.2020.06.001. Epub 2020 Jun 8. PMID 32659654
- [Background] Rush BK, Kim L, Savinoff S, Watson M, Strom L. Ask the Patient: Goals for Functional seizure treatment. Epilepsy Behav. 2024 Dec;161:110141. doi: 10.1016/j.yebeh.2024.110141. Epub 2024 Nov 13. PMID 39541741
- [Background] Goldstein LH, Robinson EJ, Chalder T, Reuber M, Medford N, Stone J, Carson A, Moore M, Landau S. Six-month outcomes of the CODES randomised controlled trial of cognitive behavioural therapy for dissociative seizures: A secondary analysis. Seizure. 2022 Mar;96:128-136. doi: 10.1016/j.seizure.2022.01.016. Epub 2022 Jan 25. PMID 35228117
- [Background] Goldstein LH, Robinson EJ, Mellers JDC, Stone J, Carson A, Reuber M, Medford N, McCrone P, Murray J, Richardson MP, Pilecka I, Eastwood C, Moore M, Mosweu I, Perdue I, Landau S, Chalder T; CODES study group. Cognitive behavioural therapy for adults with dissociative seizures (CODES): a pragmatic, multicentre, randomised controlled trial. Lancet Psychiatry. 2020 Jun;7(6):491-505. doi: 10.1016/S2215-0366(20)30128-0. Epub 2020 May 20. PMID 32445688
- [Background] Dworetzky BA. Neglected patients, few treatments, and minimal evidence: the updated cochrane review on psychological and behavioral treatments for nonepileptic seizures. Epilepsy Curr. 2014 Nov-Dec;14(6):329-31. doi: 10.5698/1535-7597-14.6.329. No abstract available. PMID 25678863
- [Background] Goldstein LH, Chalder T, Chigwedere C, Khondoker MR, Moriarty J, Toone BK, Mellers JD. Cognitive-behavioral therapy for psychogenic nonepileptic seizures: a pilot RCT. Neurology. 2010 Jun 15;74(24):1986-94. doi: 10.1212/WNL.0b013e3181e39658. PMID 20548043
- [Background] Stephen CD, Fung V, Lungu CI, Espay AJ. Assessment of Emergency Department and Inpatient Use and Costs in Adult and Pediatric Functional Neurological Disorders. JAMA Neurol. 2021 Jan 1;78(1):88-101. doi: 10.1001/jamaneurol.2020.3753. PMID 33104173
- [Background] Reuber M, Elger CE. Psychogenic nonepileptic seizures: review and update. Epilepsy Behav. 2003 Jun;4(3):205-16. doi: 10.1016/s1525-5050(03)00104-5. PMID 12791321
- [Background] Kerr WT, Zhang X, Hill CE, Janio EA, Chau AM, Braesch CT, Le JM, Hori JM, Patel AB, Allas CH, Karimi AH, Dubey I, Sreenivasan SS, Gallardo NL, Bauirjan J, Hwang ES, Davis EC, D'Ambrosio SR, Al Banna M, Cho AY, Dewar SR, Engel J Jr, Feusner JD, Stern JM. Factors associated with delay to video-EEG in dissociative seizures. Seizure. 2021 Mar;86:155-160. doi: 10.1016/j.seizure.2021.02.018. Epub 2021 Feb 15. PMID 33621828
- [Background] Kerr WT, Janio EA, Le JM, Hori JM, Patel AB, Gallardo NL, Bauirjan J, Chau AM, D'Ambrosio SR, Cho AY, Engel J Jr, Cohen MS, Stern JM. Diagnostic delay in psychogenic seizures and the association with anti-seizure medication trials. Seizure. 2016 Aug;40:123-6. doi: 10.1016/j.seizure.2016.06.015. Epub 2016 Jun 23. PMID 27398686
- [Background] LaFrance WC Jr, Baker GA, Duncan R, Goldstein LH, Reuber M. Minimum requirements for the diagnosis of psychogenic nonepileptic seizures: a staged approach: a report from the International League Against Epilepsy Nonepileptic Seizures Task Force. Epilepsia. 2013 Nov;54(11):2005-18. doi: 10.1111/epi.12356. Epub 2013 Sep 20. PMID 24111933
- [Background] Devinsky O, Gazzola D, LaFrance WC Jr. Differentiating between nonepileptic and epileptic seizures. Nat Rev Neurol. 2011 Apr;7(4):210-20. doi: 10.1038/nrneurol.2011.24. Epub 2011 Mar 8. PMID 21386814